CLINICAL TRIAL: NCT00104871
Title: A Phase II Study of Bortezomib in Metastatic Papillary Thyroid Carcinoma or Follicular Thyroid Carcinoma
Brief Title: Bortezomib in Treating Patients With Metastatic Thyroid Cancer That Did Not Respond to Radioactive Iodine Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00045; 2004-0059 (Other: UT MD Anderson Cancer Center); N01CM62202 (NIH); N01CM62203 (NIH); N01CM17003 (NIH); CDR0000415376 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Insular Thyroid Cancer; Recurrent Thyroid Cancer; Stage II Follicular Thyroid Cancer; Stage II Papillary Thyroid Cancer; Stage IV Follicular Thyroid Cancer; Stage IV Papillary Thyroid Cancer
Keywords: National Thyroid Cancer Treatment Cooperative Study Group; NTCTCSG; bortezomib; velcade; metastatic differentiated thyroid carcinoma; Differentiated thyroid carcinoma; follicular epithelial thyroid cells; papillary; oxyphilic cell; Hurthle cell; insular cell; columnar cell; tall cell
MeSH Terms: conditions — Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib (Experimental): Bortezomib 1.3 mg/m^2 intravenous (IV) at over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for at least 4 courses.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Administered IV at the dose of 1.3 mg/m^2 on a twice-weekly schedule for 2 consecutive weeks on days 1, 4, 8, and 11, followed by a 10 day rest period on days 12-21 (one cycle). In the absence of clinical progression, treatment continued for a minimum of 4 treatment cycles (or 12 weeks).
  Other Names: LDP 341; MLN341; VELCADE

SUMMARY:
This phase II trial is studying how well bortezomib works in treating patients with metastatic thyroid cancer that did not respond to radioactive iodine therapy. Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the efficacy of bortezomib, in terms of tumor response rate, in patients with metastatic papillary or follicular thyroid cancer unresponsive to prior radioiodine therapy.

SECONDARY OBJECTIVE:

I. Determine the clinical activity of this drug, in terms of progression-free survival, in patients treated with this drug.

OUTLINE: This is an open-label, multicenter study. Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for at least 4 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* The Eastern Cooperative Oncology Group (ECOG) 0-2 OR Karnofsky 60-100%
* Platelet count >= 100,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* White Blood Count (WBC) >= 3,000/mm^3
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) =< 2.5 times upper limit of normal
* Bilirubin normal
* No symptomatic congestive heart failure
* Creatinine normal OR creatinine clearance >= 60 mL/min
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* At least 4 weeks since prior chemotherapy
* No more than 2 prior chemotherapy regimens
* At least 6 months since prior external beam radiotherapy for locoregional disease in the thyroid bed or to the cervical or upper mediastinal lymph nodes (dose =< 6,000 cGy)
* At least 6 months since prior radioiodine therapy
* No prior external radiotherapy to the measured tumor
* Prior thyroidectomy allowed
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* Unresponsive to prior radioiodine therapy
* Histologically confirmed differentiated thyroid cancer-papillary or follicular type, including, but not limited to, any of the following variants: hurthle cell (oxyphilic), insular, columnar cell, tall cell
* Metastatic disease
* At least 1 unidimensionally measurable lesion >= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan
* No prior radiotherapy to the only measurable lesion
* No radioiodine uptake in the measured metastatic tumor by radioiodine scan (Note: Must have had >= 1 radioiodine scan since the last radioiodine treatment)
* No known brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-12; Primary Completion 2010-05 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Sherman, Principal Investigator — M.D. Anderson Cancer Center
Locations (9):
- United States (9):
  - University of Colorado at Denver Health Sciences Center, Aurora, Colorado
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Harvard Cancer Center, Boston, Massachusetts
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: The University of Texas MD Anderson Cancer Center official website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 2004 to April 2010. Recruitment done in medical clinics.
Pre-assignment Details: Of the 24 participants enrolled, two participants were not eligible and excluded from the study.
Period: Overall Study
Arm/Group | Bortezomib
Started | 22
Completed | 21
Not Completed | 1
Not completed — Not evaluable | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 62 [36 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response Rate Assessed by RECIST
Description: Response Rate calculated as number of participants with Complete or Partial Response divided by total participants. Baseline scan and confirmatory scans obtained 6 weeks following initial documentation of objective response using Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >30% decrease in sum longest diameter (LD) of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Baseline to 12 weeks
Population: Two participants were not evaluable for response.
Measure: Number; unit: participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 20
participants | 0

2. Primary Outcome: Participant Tumor Response Assessed by RECIST
Description: Baseline scan and confirmatory scans obtained 6 weeks following initial documentation of objective response using Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >30% decrease in sum longest diameter (LD) of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Baseline to 12 weeks (minimum of 4 treatment cycles (or 12 weeks))
Population: Two participants were not evaluable for response.
Measure: Number; unit: participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 20
participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 11
  Progressive Disease | 9

3. Secondary Outcome: Progression-free Survival Assessed by RECIST
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: At 6 months
Population: Two participants were not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 20
Participants | 4

ADVERSE EVENTS:
Time Frame: Participants followed for duration of treatment time to disease progression. Overall study period was from January 20, 2005 to May 14, 2010.
Arm/Group | Bortezomib
Serious Adverse Events (participants affected / at risk) | 17/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib (N=22)
Abdominal pain (General disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Ataxia (Nervous system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bronchial infection (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dysphasia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fatigue (General disorders) | 4
Fracture (Musculoskeletal and connective tissue disorders) | 1 — Hip Fracture
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Heart failure (Cardiac disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Insomnia (Psychiatric disorders) | 1
Investigation: Hypoalbuminemia (Investigations) | 1
Lung infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neuralgia (Nervous system disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Weight loss (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib (N=22)
Abdominal pain (Gastrointestinal disorders) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 2
Anemia (Blood and lymphatic system disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 7
Anxiety (Psychiatric disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1
Blood bilirubin increased (Investigations) | 1
Blurred vision (Eye disorders) | 1
Body odor (Skin and subcutaneous tissue disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 2
Cognitive disturbance (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Conjunctivitis (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Creatinine increased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 9
Dizziness (Nervous system disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Edema face (General disorders) | 2
Edema limbs (General disorders) | 3
Edema trunk (General disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Extrapyramidal disorder (Nervous system disorders) | 1
Eye disorders - (Other) (Eye disorders) | 2 — Scleral redness, Visual Changes
Eye infection (Infections and infestations) | 2
Eyelid function disorder (Eye disorders) | 1
Fatigue (General disorders) | 17
Fever (Investigations) | 1
Flashing Lights (Eye disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1 — Compression Fracture
Gastrointestinal disorders (Gastrointestinal disorders) | 1 — Gas
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 6
Hemorrhoids (Gastrointestinal disorders) | 1
Hot flashes (Reproductive system and breast disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hypotension (Vascular disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Infections and infestations - (Other) (Infections and infestations) | 1 — Upper Respiratory Tract
Injection site reaction (General disorders) | 1
Insomnia (Psychiatric disorders) | 6
Investigations - (Other) (Investigations) | 3 — ELEVATED lactate dehydrogenase (LDH or LD), ELEVATED blood urea nitrogen (BUN), Thrombocytopenia
Lymphocyte count decreased (Investigations) | 6
Nausea (Gastrointestinal disorders) | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 2
Non-cardiac chest pain (General disorders) | 1
Oral pain (Gastrointestinal disorders) | 1 — Mouth Soreness, Canker Sore
Pain, Body (General disorders) | 2
Pain, Knee (Musculoskeletal and connective tissue disorders) | 1
Pain, Dermis (Skin and subcutaneous tissue disorders) | 1
Gallbladder pain (Hepatobiliary disorders) | 1
Palpitations (Cardiac disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 8
Platelet count decreased (Investigations) | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Psychosis (Psychiatric disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9
Rhinitis infective (Infections and infestations) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2
Stomach pain (Gastrointestinal disorders) | 1
Testicular pain (Reproductive system and breast disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Uveitis (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Weight loss (Investigations) | 6
White blood cell decreased (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less